CLINICAL TRIAL: NCT05082428
Title: Retrospective Non-interventional Multicenter Patient Chart Data Study on Tofacitinib Realworld Experience in Ulcerative Colitis in Finland (FinTofUC)
Brief Title: This Study is to Describe and Evaluate Patients in Finland Treated With Tofacitinib for the Treatment of Ulcerative Colitis Using Real World Data.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921390; FinTofUC (Other: Alias Study Number)
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Tofacitinib: Patients treated with tofacitinib for ulcerative colitis in Finland.

SUMMARY:
The aim of this study is to describe and evaluate clinical outcomes, treatment lines, and to identify the key characteristics of the patients treated with tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Xeljanz (tofacitinib) usage for ulcerative colitis
* Diagnosis of ulcerative colitis (ICD-10: K51.0, K51.1, K51.2, K51.3, K51.5, K51.8, K51.9) between January 2010 and December 2021 (incident or prevalent).

Exclusion Criteria:

* Age < 18 years at the start of tofacitinib use
* Use of tofacitinib before reimbursement (1.3.2019)
* < 8 weeks of treatment with tofacitinib at the start of data mining
* History of panproctocolectomy, IPAA or ileostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective non-interventional multicenter patient chart review study, collecting real world data from 21 Finnish hospital district databases and for whom data is available.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Molander P, Kosunen M, Eronen H, Tillonen J, Karajamaki A, Heikkinen M, Punkkinen J, Mattila R, Toppila I, Holsa O, Kalpala K, Henrohn D, Af Bjorkesten CG. Tofacitinib real-world experience in ulcerative colitis in Finland (FinTofUC): a retrospective non-interventional multicenter patient chart data study. Scand J Gastroenterol. 2024 Apr;59(4):425-432. doi: 10.1080/00365521.2023.2298361. Epub 2023 Dec 29. PMID 38156792
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of ulcerative colitis (UC) between January 2010 and December 2021 and who initiated tofacitinib across Finland were included in this retrospective chart study. Data was collected from patient registers and charts in Finland. Index date was considered as date of initiation of tofacitinib treatment for ulcerative colitis. Data was collected and analyzed over 5 months in this retrospective study.
Groups:
- Tofacitinib: Participants diagnosed with UC between January 2010 and December 2021 and who initiated tofacitinib were included.
Period: Overall Study
Arm/Group | Tofacitinib
Started | 252
Completed | 252
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants for whom data was collected and analyzed were included.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at index (date of initiation of tofacitinib treatment for ulcerative colitis)
  Years | 38.94 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 175
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kilograms] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  Kilograms
    number analyzed (Participants) | 85
    (all) | 81.54 (19.47)
Height [Mean (Standard Deviation); unit: Centimeters] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  Centimeters
    number analyzed (Participants) | 54
    (all) | 174.63 (8.33)
Smoking status [Count of Participants; unit: Participants] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  Participants
    number analyzed (Participants) | 220
    Current | 16
    Ex-smoker | 43
    Non-smoker | 161
Body Mass Index [Mean (Standard Deviation); unit: Kilogram per meter square] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  Kilogram per meter square
    number analyzed (Participants) | 209
    (all) | 26.5 (5.8)
Absolute Value of Plasma C-reactive Protein at Baseline [Mean (Standard Deviation); unit: Milligrams per liter] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  Milligrams per liter
    number analyzed (Participants) | 199
    (all) | 8.97 (11.93)
Absolute Values of Blood leukocytes, lymphocytes, neutrophiles, and thrombocytes [Mean (Standard Deviation); unit: 10^9 cells per liter] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  10^9 cells per liter
    Blood leukocytes: number analyzed (Participants) | 213
    Blood leukocytes | 10.86 (32.06)
    Blood lymphocytes: number analyzed (Participants) | 149
    Blood lymphocytes | 2.08 (0.95)
    Blood neutrophiles: number analyzed (Participants) | 146
    Blood neutrophiles | 5.78 (3.85)
    Blood thrombocytes: number analyzed (Participants) | 210
    Blood thrombocytes | 336.55 (115.87)
Absolute Value of Fecal Calprotectin at Index [Mean (Standard Deviation); unit: Milligrams per kilogram] — Population: 'Number Analyzed' signifies participants evaluable for specified rows.
  Milligrams per kilogram
    number analyzed (Participants) | 189
    (all) | 1907.43 (1716.94)

OUTCOME MEASURES:

1. Primary Outcome: Age at the Time of Diagnosis
Description: Participant's age at the time of ulcerative colitis diagnosis was presented in this outcome measure. Index was considered as date of initiation of tofacitinib treatment for ulcerative colitis.
Time Frame: At diagnosis (anytime between Jan 2010 and Dec-2021, approximately 12 years (from data collected and analyzed retrospectively over 5 months)
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Years | 31.08 (13.02)

2. Primary Outcome: Duration of Ulcerative Colitis
Description: Duration of ulcerative colitis was presented in this outcome measure. Index was considered as date of initiation of tofacitinib treatment for ulcerative colitis.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Years | 7.91 (7.79)

3. Primary Outcome: Number of Participants With Extent of Colonic Involvement According to the Montreal Classification
Description: Montreal classification was used to classify UC based on extent of inflammation. Three subgroups of UC were: E1= ulcerative proctitis: involvement limited to rectum i.e, proximal extent of inflammation is distal to rectosigmoid junction, E2= left sided, distal colitis: involvement limited to portion of colorectum distal to splenic flexure and E3= extensive UC (pancolitis): involvement extends proximal to the splenic flexure. Index was considered as date of initiation of tofacitinib treatment for UC.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: All eligible participants for whom data was collected and analyzed were included. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  E1 | 5
  E2 | 67
  E3 | 180

4. Primary Outcome: Mayo Score at Initiation of Tofacitinib
Description: Mayo score was composed of four components: rectal bleeding, stool frequency, physician (doctors) assessment of disease activity, and endoscopy findings. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity. Index was considered as date of initiation of tofacitinib treatment for ulcerative colitis. Mayo scores and sub-scores have been collected by doctors independently as part of standard of care.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: All eligible participants for whom data was collected and analyzed were included. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 80
Units on a scale | 7.45 (2.43)

5. Primary Outcome: Partial Mayo Score at Initiation of Tofacitinib
Description: Partial Mayo score consisted of 3 components: rectal bleeding, stool frequency, and physician (doctors) assessment of disease activity. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity. Index was considered as date of initiation of tofacitinib treatment for ulcerative colitis. Partial Mayo scores and sub-scores have been collected by doctors independently as part of standard of care.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Tofacitinib
Number analyzed (Participants) | 203
Years | 4.75 (2.06)

6. Primary Outcome: Number of Participants According to Endoscopic Findings Based on Histology
Description: Endoscopic findings were graded from 0 to 3 where 0 = Normal or inactive disease (Normal vascular pattern with arborization of capillaries clearly defined, or with blurring or patchy loss of capillary margins), 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration). Index was considered as date of initiation of tofacitinib treatment for ulcerative colitis.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 85
Participants
  Active disease | NA — Any participant groups of <5 participants cannot be exported from the Finnish Health and Social Data Permit Authority (Findata) servers. Any information which enables to calculate <5 participant group information based on information from another participants group will not be presented.
  Inactive disease | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Normal histology | 0

7. Primary Outcome: Number of Participants According to Endoscopic Sub Score Based on Mayo Score
Description: Endoscopic findings were graded from 0 to 3 where 0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 3 = Severe disease (spontaneous bleeding, ulceration). Mayo score was composed of four components: rectal bleeding, stool frequency, physician assessment of disease activity and endoscopy findings. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity. Index was considered as date of initiation of tofacitinib treatment for ulcerative colitis.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 88
Participants
  Sub score 1 | 10
  Sub score 2 | 42
  Sub score 3 | 36

8. Secondary Outcome: Percentage of Participants Who Received Tofacitinib at Week 8, Week 16, Week 24 and Week 52
Description: Percentage of participants who received tofacitinib is presented in this outcome measure.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8 | 91.67
  Week 16 | 80.16
  Week 24 | 71.03
  Week 52: number analyzed (Participants) | 212
  Week 52 | 54.72

9. Secondary Outcome: Percentage of Participants With Clinical Remission Based on Full Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical remission in participants was defined as a full Mayo score of less than or equal to (<=) 2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings. Each subscore ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score which ranged from 0 to 12, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: All eligible participants for whom data was collected and analyzed were included. 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 91
  Week 8 | 5.49
  Week 16: number analyzed (Participants) | 105
  Week 16 | 9.52
  Week 24: number analyzed (Participants) | 116
  Week 24 | 14.66
  Week 52: number analyzed (Participants) | 129
  Week 52 | 20.16

10. Secondary Outcome: Percentage of Participants With Clinical Remission Based on Partial Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical remission in participants was defined as a partial Mayo score of less than 2 points with rectal bleeding sub-score of 0. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 219
  Week 8 | 28.77
  Week 16: number analyzed (Participants) | 230
  Week 16 | 36.52
  Week 24: number analyzed (Participants) | 232
  Week 24 | 34.91
  Week 52: number analyzed (Participants) | 202
  Week 52 | 33.66

11. Secondary Outcome: Percentage of Participants With Clinical Response Based on Full Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical response in participants was defined as a full Mayo score decrease of greater than or equal (>=) to 3 points and a decrease of >=30 percent (%) from baseline, with a decrease of >=1 point on the rectal bleeding sub score or an absolute rectal bleeding score of less than equal to (<=)1. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 80
  Week 8 | 32.5
  Week 16: number analyzed (Participants) | 80
  Week 16 | 38.75
  Week 24: number analyzed (Participants) | 80
  Week 24 | 35
  Week 52: number analyzed (Participants) | 69
  Week 52 | 26.09

12. Secondary Outcome: Percentage of Participants With Clinical Response Based on Partial Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical response in participants was defined as a partial Mayo score decrease of >=2 points and reduction of at least 25% in partial Mayo score from baseline with an accompanying decrease in rectal bleeding sub score of >=1 point or absolute rectal bleeding sub score of <=1. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 203
  Week 8 | 37.44
  Week 16: number analyzed (Participants) | 203
  Week 16 | 44.83
  Week 24: number analyzed (Participants) | 203
  Week 24 | 42.86
  Week 52: number analyzed (Participants) | 174
  Week 52 | 33.33

13. Secondary Outcome: Percentage of Participants With Steroid-free Clinical Remission for All Participants Based on Full Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical remission in participants was defined as a full Mayo score of <=2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 91
  Week 8 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 16: number analyzed (Participants) | 105
  Week 16 | 6.67
  Week 24: number analyzed (Participants) | 116
  Week 24 | 12.93
  Week 52: number analyzed (Participants) | 129
  Week 52 | 19.38

14. Secondary Outcome: Percentage of Participants With Steroid-free Clinical Remission for All Participants Based on Partial Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical remission in participants was defined as a partial Mayo score of less than 2 points with rectal bleeding sub-score of 0. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity. Steroid-free clinical remission was defined for participants who were treated with corticosteroids at baseline and did not require any corticosteroid treatment during the period >=4 weeks prior to the visit.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 219
  Week 8 | 10.5
  Week 16: number analyzed (Participants) | 230
  Week 16 | 31.74
  Week 24: number analyzed (Participants) | 232
  Week 24 | 30.17
  Week 52: number analyzed (Participants) | 202
  Week 52 | 31.19

15. Secondary Outcome: Percentage of Participants According to Time to Response Based on Full or Partial Mayo Score at 1, 2, 3, 6, 12, 24, 36 Months
Description: Time to clinical response was analyzed using a competing risk time-to-event model, where clinical response and drug discontinuation were assessed. Clinical response in participants was defined as full Mayo score decrease of >=3 points & decrease of >=30% from baseline, with decrease of >=1 point on rectal bleeding sub score or absolute rectal bleeding score of <=1. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, & endoscopy findings. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). Sub scores were summed up to give total score range: 0 to 12, Partial Mayo score consisted of 3 components without endoscopy findings. Each graded from 0 to 3, sub scores were summed up to give total score range: 0 to 9.Higher scores indicated higher disease severity.
Time Frame: At 1, 2, 3, 6, 12, 24 and 36 months
Population: All eligible participants for whom data was collected and analyzed were included. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies maximum participants evaluable at specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 203
Percentage of participants
  1 month | 15.3 [11.0 to 21.1]
  2 months | 45.8 [39.4 to 53.2]
  3 months | 56.2 [49.7 to 63.4]
  6 months | 67.0 [60.8 to 73.8]
  12 months: number analyzed (Participants) | 189
  12 months | 70.5 [64.5 to 77.1]
  24 months: number analyzed (Participants) | 80
  24 months | 72.2 [66.1 to 78.8]
  36 months: number analyzed (Participants) | 57
  36 months | 75.2 [68.8 to 82.2]

16. Secondary Outcome: Percentage of Participants With Fecal (F)-Calprotectin Reduction of >=50% at Week 8, Week 16, Week 24 and Week 52
Description: F-calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Percentage of participants with F-calprotectin reduction of >=50% from baseline at Week 8, Week 16, Week 24 and Week 52 is presented.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 189
  Week 8 | 29.1
  Week 16: number analyzed (Participants) | 189
  Week 16 | 46.56
  Week 24: number analyzed (Participants) | 189
  Week 24 | 45.5
  Week 52: number analyzed (Participants) | 158
  Week 52 | 37.34

17. Secondary Outcome: Percentage of Participants With F-calprotectin Reduction of >=75% at Week 8, Week 16, Week 24 and Week 52
Description: F-calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Percentage of participants with F-calprotectin reduction of >=75% compared to baseline at Week 8, Week 16, Week 24 and Week 52 is presented.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 189
  Week 8 | 20.63
  Week 16: number analyzed (Participants) | 189
  Week 16 | 36.51
  Week 24: number analyzed (Participants) | 189
  Week 24 | 37.04
  Week 52: number analyzed (Participants) | 158
  Week 52 | 32.28

18. Secondary Outcome: Percentage of Participants With F-calprotectin Reduction of >=90% at Week 8, Week 16, Week 24 and Week 52
Description: F-calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Percentage of participants with F-calprotectin reduction of >=90% compared to baseline at Week 8, Week 16, Week 24 and Week 52 is presented.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 189
  Week 8 | 12.17
  Week 16: number analyzed (Participants) | 189
  Week 16 | 24.34
  Week 24: number analyzed (Participants) | 189
  Week 24 | 25.93
  Week 52: number analyzed (Participants) | 158
  Week 52 | 23.42

19. Secondary Outcome: Number of Participants Reaching F-calprotectin Below 250 mg/kg of Those That Had F-calprotectin Above 250 mg/kg at Baseline
Description: F-calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Percentage of participants reaching F-calprotectin below 250mg/kg at Week 8, Week 16, Week 24 and Week 52 in those participants who had F-calprotectin above 250 mg/kg at Baseline is presented.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 171
Participants
  Week 8 | 31
  Week 16 | 55
  Week 24 | 58
  Week 52 | 44

20. Secondary Outcome: Change From Baseline in F-calprotectin at Week 8, Week 16, Week 24 and Week 52 With F-Calprotectin Above 250 mg/kg at Baseline
Description: F-calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation. Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligrams per kilogram
Arm/Group | Tofacitinib
Number analyzed (Participants) | 171
Milligrams per kilogram
  Week 8 | -594.83 (1302.24)
  Week 16 | -1100.28 (1653.91)
  Week 24 | -1291.7 (1589.91)
  Week 52 | -1393.53 (1727.43)

21. Secondary Outcome: Percentage of Participants in Sustained Remission Based on Full Mayo Score From Week 8 to Week 16, Week 24, and Week 52
Description: Sustained remission in participants was defined as a full Mayo score of <=2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity.
Time Frame: From Week 8 to Week 16, Week 24, and Week 52
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 5
Percentage of Participants
  Week 8 to Week 16 | 100.0
  Week 8 to Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 8 to Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.

22. Secondary Outcome: Percentage of Participants in Sustained Remission Based on Partial Mayo Score From Week 8 to Week 16, Week 24, and Week 52
Description: Sustained remission in participants was defined as a partial score of less than 2 points with rectal bleeding sub-score of 0. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity.
Time Frame: From Week 8 to Week 16, Week 24 and Week 52
Population: All eligible participants for whom data was collected and analyzed were included. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 63
Percentage of Participants
  Week 8 to Week 16 | 84.13
  Week 8 to Week 24 | 63.49
  Week 8 to Week 52: number analyzed (Participants) | 55
  Week 8 to Week 52 | 50.91

23. Secondary Outcome: Percentage of Participants in Sustained Remission Based on Full Mayo Score From Week 16 to Week 24 and Week 52
Description: Sustained remission in participants was defined as a full Mayo score of >=2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity.
Time Frame: From Week 16 to Week 24 and Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 10
Percentage of Participants
  Week 16 to Week 24 | 90.0
  Week 16 to Week 52: number analyzed (Participants) | 8
  Week 16 to Week 52 | 75.0

24. Secondary Outcome: Percentage of Participants in Sustained Remission Based on Partial Mayo Score From Week 16 to Week 24 and Week 52
Description: as for outcome 22
Time Frame: From Week 16 to Week 24 and Week 52
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 84
Percentage of Participants
  Week 16 to Week 24 | 76.19
  Week 16 to Week 52: number analyzed (Participants) | 70
  Week 16 to Week 52 | 64.29

25. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission Based on Full Mayo Score From Week 16 to Week 24 and Week 52
Description: Clinical remission in participants was defined as a full Mayo score of <=2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity. Steroid-free clinical remission was defined as clinical remission in participants who were treated with corticosteroids at baseline and did not require any corticosteroid treatment during the period >=4 weeks prior to the visit.
Time Frame: From Week 16 to Week 24 and Week 52
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 7
Percentage of Participants
  Week 16 to Week 24 | 85.71
  Week 16 to Week 52 | 71.43

26. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission Based on Partial Mayo Score From Week 16 to Week 24 and Week 52
Description: Clinical remission in participants was defined as a partial score of less than 2 points with rectal bleeding sub-score of 0. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity. Steroid-free clinical remission was defined as clinical remission in participants who were treated with corticosteroids at baseline and did not require any corticosteroid treatment during the period >=4 weeks prior to the visit.
Time Frame: From Week 16 to Week 24 and Week 52
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 70
Percentage of Participants
  Week 16 to Week 24 | 72.6
  Week 16 to Week 52: number analyzed (Participants) | 61
  Week 16 to Week 52 | 60.66

27. Secondary Outcome: Change From Baseline in Full Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Mayo score was an instrument designed to measure disease activity of UC. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity. Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Units on a scale
  Week 8: number analyzed (Participants) | 80
  Week 8 | -1.9 (2.3)
  Week 16: number analyzed (Participants) | 80
  Week 16 | -2.39 (2.51)
  Week 24: number analyzed (Participants) | 80
  Week 24 | -2.63 (2.13)
  Week 52: number analyzed (Participants) | 69
  Week 52 | -2.66 (2.92)

28. Secondary Outcome: Change From Baseline in Partial Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity. Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Units on a scale
  Week 8: number analyzed (Participants) | 203
  Week 8 | -1.62 (2.22)
  Week 16: number analyzed (Participants) | 203
  Week 16 | -2.21 (2.32)
  Week 24: number analyzed (Participants) | 203
  Week 24 | -2.4 (2.13)
  Week 52: number analyzed (Participants) | 174
  Week 52 | -2.43 (2.61)

29. Secondary Outcome: Percentage of Participants in Sustained Endoscopic Remission, Mucosal Healing or Endoscopic Response From Week 8 to Week 16, Week 24 and Week 52
Description: Sustained endoscopic remission was defined as Mayo endoscopic sub score of 0. Mucosal healing = Mayo endoscopic sub score of 0 or 1. Endoscopic response= sub score reduction from baseline of >=1. The Mayo endoscopic sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). Higher sub scores indicated higher disease severity.
Time Frame: From Week 8 to Week 16, Week 24 and Week 52
Population: as for outcome 22
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 11
Percentage of participants
  Week 8 to Week 16 | 100
  Week 8 to Week 24 | 100
  Week 8 to Week 52: number analyzed (Participants) | 10
  Week 8 to Week 52 | 50

30. Secondary Outcome: Percentage of Participants With Physician Assessed Histological Remission at Week 8, Week 16, Week 24 and Week 52
Description: Physician assessed histological remission was defined as inactive disease or normal histology. Inactive disease was characterized by marked architectural abnormalities in the absence of active inflammation.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 93
  Week 8 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 16: number analyzed (Participants) | 102
  Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 24: number analyzed (Participants) | 113
  Week 24 | 6.19
  Week 52: number analyzed (Participants) | 122
  Week 52 | 11.48

31. Secondary Outcome: Change From Baseline in Histology Assessment at Week 8, Week 16, Week 24 and Week 52
Description: Histology assessment was categorized as, 1= inactive disease or normal histology and 2 = active disease. Inactive disease was characterized by marked architectural abnormalities in the absence of active inflammation. Active disease was characterized by absence of active inflammation. Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Units on a scale
  Week 8: number analyzed (Participants) | 85
  Week 8 | 0 (0)
  Week 16: number analyzed (Participants) | 85
  Week 16 | -0.01 (0.12)
  Week 24: number analyzed (Participants) | 85
  Week 24 | -0.02 (0.13)
  Week 52: number analyzed (Participants) | 73
  Week 52 | -0.18 (0.52)

32. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission for All Participants Based on Full Mayo Score and Endoscopic Remission, Mucosal Healing or Endoscopic Response From Week 8 to Week 16, Week 24 and Week 52
Description: Sustained endoscopic remission was defined as Mayo endoscopic sub score of 0. Mucosal healing was defined by Mayo endoscopic sub score of 0 or 1. Endoscopic response was defined as sub score reduction from baseline of >=1. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity. Steroid-free clinical remission was defined as clinical remission in participants who were treated with corticosteroids at baseline and did not require any corticosteroid treatment during the period >=4 weeks prior to the visit.
Time Frame: From Week 8 to Week 16, Week 24 and Week 52
Population: All eligible participants for whom data was collected and analyzed were included. "Overall Number of Participants Analyzed" signifies maximum number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 4
Percentage of participants
  Week 8 to Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 8 to Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 8 to Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.

33. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission for All Participants Based on Partial Mayo Score and Endoscopic Remission, Mucosal Healing or Endoscopic Response From Week 8 to Week 16, Week 24 and Week 52
Description: Sustained endoscopic remission was defined as Mayo endoscopic sub score of 0. Mucosal healing was defined by Mayo endoscopic sub score of 0 or 1. Endoscopic response was defined as sub score reduction from baseline of >=1. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity. Steroid-free clinical remission was defined as participants who were treated with corticosteroids at baseline and did not require any corticosteroid treatment during the period >=4 weeks prior to the visit.
Time Frame: From Week 8 to Week 16, Week 24 and Week 52
Population: as for outcome 32
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 4
Percentage of participants
  Week 8 to Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 8 to Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 8 to Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.

34. Secondary Outcome: Number of Participants With Clinical Remission Based on Full Mayo Score According to Montreal Classification at Week 8, Week 16, Week 24, and Week 52
Description: Montreal classification was system used to classify UC based on the extent of inflammation. Three subgroups of UC were defined by extent of colonic involvement: E1= ulcerative proctitis: involvement limited to the rectum i.e, proximal extent of inflammation is distal to rectosigmoid junction, E2= left sided UC also known as distal colitis: involvement limited to portion of colorectum distal to the splenic flexure, E3= extensive UC (pancolitis): involvement extents proximal to splenic flexure. Clinical remission: full Mayo score of <=2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, & endoscopy findings, each sub score ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give total score range of 0 to 12. Higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24, and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  E1 ulcerative proctitis, Week 8: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 8 | 0
  E1 ulcerative proctitis, Week 16: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 16 | 0
  E1 ulcerative proctitis, Week 24: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 24 | 0
  E1 ulcerative proctitis, Week 52: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E2 left-sided UC, Week 8: number analyzed (Participants) | 67
  E2 left-sided UC, Week 8 | 0
  E2 left-sided UC, Week 16: number analyzed (Participants) | 67
  E2 left-sided UC, Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E2 left-sided UC, Week 24: number analyzed (Participants) | 67
  E2 left-sided UC, Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E2 left-sided UC, Week 52: number analyzed (Participants) | 53
  E2 left-sided UC, Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E3 extensive UC, Week 8: number analyzed (Participants) | 180
  E3 extensive UC, Week 8 | 5
  E3 extensive UC, Week 16: number analyzed (Participants) | 180
  E3 extensive UC, Week 16 | 8
  E3 extensive UC, Week 24: number analyzed (Participants) | 180
  E3 extensive UC, Week 24 | 15
  E3 extensive UC, Week 52: number analyzed (Participants) | 155
  E3 extensive UC, Week 52 | 22

35. Secondary Outcome: Number of Participants With Clinical Remission Based on Partial Mayo Score According to Montreal Classification at Week 8, Week 16, Week 24, and Week 52
Description: Montreal Classification was system used to classify UC based on the extent of inflammation. Three subgroups of UC were defined by extent of colonic involvement: E1= ulcerative proctitis: involvement limited to the rectum i.e, proximal extent of inflammation is distal to rectosigmoid junction, E2= left sided UC also known as distal colitis: involvement limited to portion of colorectum distal to the splenic flexure, E3= extensive UC (pancolitis): involvement extents proximal to splenic flexure. Clinical remission: partial score of less than 2 points with rectal bleeding sub-score of 0. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24, and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  E1 ulcerative proctitis, Week 8: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 8 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 16: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 24: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 52: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E2 left-sided UC, Week 8: number analyzed (Participants) | 67
  E2 left-sided UC, Week 8 | 12
  E2 left-sided UC, Week 16: number analyzed (Participants) | 67
  E2 left-sided UC, Week 16 | 21
  E2 left-sided UC, Week 24: number analyzed (Participants) | 67
  E2 left-sided UC, Week 24 | 17
  E2 left-sided UC, Week 52: number analyzed (Participants) | 53
  E2 left-sided UC, Week 52 | 16
  E3 extensive UC, Week 8: number analyzed (Participants) | 180
  E3 extensive UC, Week 8 | 50
  E3 extensive UC, Week 16: number analyzed (Participants) | 180
  E3 extensive UC, Week 16 | 62
  E3 extensive UC, Week 24: number analyzed (Participants) | 180
  E3 extensive UC, Week 24 | 63
  E3 extensive UC, Week 52: number analyzed (Participants) | 155
  E3 extensive UC, Week 52 | 52

36. Secondary Outcome: Number of Participants With Clinical Response Based on Full Mayo Score According to Montreal Classification at Week 8, Week 16, Week 24, and Week 52
Description: Montreal Classification was used to classify ulcerative colitis (UC) based on extent of inflammation. Three subgroups of UC were: E1= ulcerative proctitis: involvement limited to rectum i.e, proximal extent of inflammation is distal to rectosigmoid junction, E2= left sided, distal colitis: involvement limited to portion of colorectum distal to splenic flexure and E3= extensive UC (pancolitis): involvement extends proximal to the splenic flexure. Clinical response: full Mayo score decrease of >= 3 points & decrease of >=30% from baseline, with decrease of >=1 point on rectal bleeding sub score or an absolute rectal bleeding score of less than equal to (<=)1. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12. Higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24, and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  E1 ulcerative proctitis, Week 8: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 8 | 0
  E1 ulcerative proctitis, Week 16: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 24: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 52: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E2 left-sided UC, Week 8: number analyzed (Participants) | 67
  E2 left-sided UC, Week 8 | 8
  E2 left-sided UC, Week 16: number analyzed (Participants) | 67
  E2 left-sided UC, Week 16 | 11
  E2 left-sided UC, Week 24: number analyzed (Participants) | 67
  E2 left-sided UC, Week 24 | 10
  E2 left-sided UC, Week 52: number analyzed (Participants) | 53
  E2 left-sided UC, Week 52 | 6
  E3 extensive UC, Week 8: number analyzed (Participants) | 180
  E3 extensive UC, Week 8 | 18
  E3 extensive UC, Week 16: number analyzed (Participants) | 180
  E3 extensive UC, Week 16 | 19
  E3 extensive UC, Week 24: number analyzed (Participants) | 180
  E3 extensive UC, Week 24 | 17
  E3 extensive UC, Week 52: number analyzed (Participants) | 155
  E3 extensive UC, Week 52 | 11

37. Secondary Outcome: Number of Participants With Clinical Response Based on Partial Mayo Score According to Montreal Classification at Week 8, Week 16, Week 24, and Week 52
Description: Montreal Classification was used to classify ulcerative colitis (UC) based on extent of inflammation. Three subgroups of UC were: E1= ulcerative proctitis: involvement limited to rectum i.e, proximal extent of inflammation is distal to rectosigmoid junction, E2= left sided, distal colitis: involvement limited to portion of colorectum distal to splenic flexure and E3= extensive UC (pancolitis): involvement extends proximal to the splenic flexure. Clinical response: full Mayo score decrease of >=3 points and decrease of >=30% from baseline, with a decrease of >=1 point on rectal bleeding sub score or an absolute rectal bleeding score of less than equal to (<=)1. Partial Mayo score consisted of 3 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity. Each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 9, where higher scores indicated higher disease severity.
Time Frame: Week 8, Week 16, Week 24, and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  E1 ulcerative proctitis, Week 8: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 8 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 16: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 24: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E1 ulcerative proctitis, Week 52: number analyzed (Participants) | 5
  E1 ulcerative proctitis, Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  E2 left-sided UC, Week 8: number analyzed (Participants) | 67
  E2 left-sided UC, Week 8 | 20
  E2 left-sided UC, Week 16: number analyzed (Participants) | 67
  E2 left-sided UC, Week 16 | 24
  E2 left-sided UC, Week 24: number analyzed (Participants) | 67
  E2 left-sided UC, Week 24 | 24
  E2 left-sided UC, Week 52: number analyzed (Participants) | 53
  E2 left-sided UC, Week 52 | 14
  E3 extensive UC, Week 8: number analyzed (Participants) | 180
  E3 extensive UC, Week 8 | 55
  E3 extensive UC, Week 16: number analyzed (Participants) | 180
  E3 extensive UC, Week 16 | 65
  E3 extensive UC, Week 24: number analyzed (Participants) | 180
  E3 extensive UC, Week 24 | 61
  E3 extensive UC, Week 52: number analyzed (Participants) | 155
  E3 extensive UC, Week 52 | 43

38. Secondary Outcome: Percentage of Participants With Corticosteroid Tapering at Week 8, Week 16, Week 24 and Week 52
Description: Percentage of participants with corticosteroid tapering response was collected as Yes or No based on latest available data.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants | NA — As this was a retrospective study, doses were not recorded in patient registry

39. Secondary Outcome: Tapering Rate
Description: Corticosteroid tapering rate is reported in this outcome measure.
Time Frame: Up to Week 52
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Mean (Standard Deviation); unit: Milligram per day
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Milligram per day | NA (NA) — As this was a retrospective study, doses were not recorded in patient registry

40. Secondary Outcome: Corticosteroid Tapering Dose
Time Frame: Up to Week 52
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Milligrams | NA (NA) — As this was a retrospective study, doses were not recorded in patient registry

41. Secondary Outcome: Percentage of Participants With Improvement in Stool Frequency Sub Score of 1 or More Points at Week 8, Week 16, Week 24 and Week 52
Description: Stool frequency sub score ranged from 0 to 3, where, 0 = Normal, 1 = 1 to 2 stools per day more than normal, 2 = 3 to 4 stools per day more than normal, 3 = 5 or more stools per day than normal. Percentage of participants with improvement in stool frequency sub score of 1 or more points is presented.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 213
  Week 8 | 38.03
  Week 16: number analyzed (Participants) | 213
  Week 16 | 45.07
  Week 24: number analyzed (Participants) | 213
  Week 24 | 41.78
  Week 52: number analyzed (Participants) | 181
  Week 52 | 32.6

42. Secondary Outcome: Change From Baseline in Stool Frequency Sub Score at Week 8, Week 16, Week 24 and Week 52
Description: Stool frequency sub score ranged from 0 to 3, where, 0 = Normal, 1 = 1 to 2 stools per day more than normal, 2 = 3 to 4 stools per day more than normal, 3 = 5 or more stools per day than normal.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: All eligible participants for whom data was collected and analyzed were included. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints. 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Units on a scale
  Week 8: number analyzed (Participants) | 213
  Week 8 | -0.62 (0.97)
  Week 16: number analyzed (Participants) | 213
  Week 16 | -0.86 (1.03)
  Week 24: number analyzed (Participants) | 213
  Week 24 | -0.97 (0.99)
  Week 52: number analyzed (Participants) | 181
  Week 52 | -1.01 (1.2)

43. Secondary Outcome: Percentage of Participants With Improvement in Rectal Bleeding Sub Score of 1 or More Points at Week 8, Week 16, Week 24 and Week 52
Description: Rectal bleeding sub scores ranged from 0 to 3, where, 0 = None, 1 = Visible blood with stool less than half the time, 2 = Visible blood with stool half of the time or more, 3 = Passing blood alone. Percentage of participants with improvement in rectal bleeding sub score of 1 or more points are presented.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of participants
  Week 8: number analyzed (Participants) | 217
  Week 8 | 28.57
  Week 16: number analyzed (Participants) | 217
  Week 16 | 29.49
  Week 24: number analyzed (Participants) | 217
  Week 24 | 28.11
  Week 52: number analyzed (Participants) | 184
  Week 52 | 22.83

44. Secondary Outcome: Change From Baseline in Rectal Bleeding Sub Score at Week 8, Week 16, Week 24 and Week 52
Description: Rectal bleeding sub scores ranged from 0 to 3, where, 0 = None, 1 = Visible blood with stool less than half the time, 2 = Visible blood with stool half of the time or more, 3 = Passing blood alone. Baseline was considered as initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Units on a scale
  Week 8: number analyzed (Participants) | 217
  Week 8 | -0.41 (0.8)
  Week 16: number analyzed (Participants) | 217
  Week 16 | -0.49 (0.91)
  Week 24: number analyzed (Participants) | 217
  Week 24 | -0.47 (0.87)
  Week 52: number analyzed (Participants) | 184
  Week 52 | -0.53 (1.02)

45. Secondary Outcome: Percentage of Participants Reaching Normal P-CRP, B-hb, B-leuk, B-Thromb, B-ly, B-Neutr and P-alb Levels at Week 8, Week 16, Week 24 and Week 52
Description: Normal values for the parameters were as follows: P-CRP: below 4 milligrams per liter (mg/L), B-hb: men: 134 to 167 grams per liter (g/L), women: 117-155 g/L, B-leuk: 3.4 to 8.2*10^9 cells/L, B-Thromb: 150 to 360*10^9 cells/L, B-ly: 1.3 to3.6*10^9 cells/L, B-Neutr: 1.5 to6.7*10^9 cells/L, P-alb: 18 to 39 years: 36 to 48 g/L, 40 to 69 years: 36 to 45 g/L, 70 years and over: 34 to 45 g/L.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of participants
  P-CRP, Week 8: number analyzed (Participants) | 227
  P-CRP, Week 8 | 67.4
  P-CRP, Week 16: number analyzed (Participants) | 245
  P-CRP, Week 16 | 61.63
  P-CRP, Week 24: number analyzed (Participants) | 247
  P-CRP, Week 24 | 57.09
  P-CRP, Week 52: number analyzed (Participants) | 211
  P-CRP, Week 52 | 44.55
  B-hb, Week 8: number analyzed (Participants) | 239
  B-hb, Week 8 | 70.29
  B-hb, Week 16: number analyzed (Participants) | 249
  B-hb, Week 16 | 63.45
  B-hb, Week 24: number analyzed (Participants) | 249
  B-hb, Week 24 | 58.23
  B-hb, Week 52: number analyzed (Participants) | 211
  B-hb, Week 52 | 48.82
  B-leuk, Week 8: number analyzed (Participants) | 237
  B-leuk, Week 8 | 59.92
  B-leuk, Week 16: number analyzed (Participants) | 247
  B-leuk, Week 16 | 60.73
  B-leuk, Week 24: number analyzed (Participants) | 247
  B-leuk, Week 24 | 53.85
  B-leuk, Week 52: number analyzed (Participants) | 209
  B-leuk, Week 52 | 43.54
  B-Thromb, Week 8: number analyzed (Participants) | 237
  B-Thromb, Week 8 | 64.98
  B-Thromb, Week 16: number analyzed (Participants) | 247
  B-Thromb, Week 16 | 59.92
  B-Thromb, Week 24: number analyzed (Participants) | 248
  B-Thromb, Week 24 | 55.65
  B-Thromb, Week 52: number analyzed (Participants) | 211
  B-Thromb, Week 52 | 43.6
  B-ly, Week 8: number analyzed (Participants) | 206
  B-ly, Week 8 | 74.76
  B-ly, Week 16: number analyzed (Participants) | 226
  B-ly, Week 16 | 67.7
  B-ly, Week 24: number analyzed (Participants) | 227
  B-ly, Week 24 | 59.03
  B-ly, Week 52: number analyzed (Participants) | 196
  B-ly, Week 52 | 45.41
  B-Neutr, Week 8: number analyzed (Participants) | 199
  B-Neutr, Week 8 | 79.9
  B-Neutr, Week 16: number analyzed (Participants) | 212
  B-Neutr, Week 16 | 72.17
  B-Neutr, Week 24: number analyzed (Participants) | 213
  B-Neutr, Week 24 | 64.79
  B-Neutr, Week 52: number analyzed (Participants) | 183
  B-Neutr, Week 52 | 48.09
  P-alb, Week 8: number analyzed (Participants) | 183
  P-alb, Week 8 | 62.3
  P-alb, Week 16: number analyzed (Participants) | 212
  P-alb, Week 16 | 57.08
  P-alb, Week 24: number analyzed (Participants) | 214
  P-alb, Week 24 | 51.4
  P-alb, Week 52: number analyzed (Participants) | 191
  P-alb, Week 52 | 45.55

46. Secondary Outcome: Change From Baseline in P-CRP Levels at Week 8, Week 16, Week 24 and Week 52
Description: Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Milligrams per liter
  Week 8: number analyzed (Participants) | 199
  Week 8 | -1.06 (10.19)
  Week 16: number analyzed (Participants) | 199
  Week 16 | -1.31 (8.49)
  Week 24: number analyzed (Participants) | 199
  Week 24 | -1.74 (8.19)
  Week 52: number analyzed (Participants) | 168
  Week 52 | -2.36 (9.91)

47. Secondary Outcome: Change From Baseline in B-hb and P-alb Levels at Week 8, Week 16, Week 24 and Week 52
Description: Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Grams per liter
  B-hb, Week 8: number analyzed (Participants) | 215
  B-hb, Week 8 | 0.71 (9.88)
  B-hb, Week 16: number analyzed (Participants) | 215
  B-hb, Week 16 | 1.19 (10.75)
  B-hb, Week 24: number analyzed (Participants) | 215
  B-hb, Week 24 | 1.11 (10.51)
  B-hb, Week 52: number analyzed (Participants) | 183
  B-hb, Week 52 | 3.77 (12.64)
  P-alb, Week 8: number analyzed (Participants) | 150
  P-alb, Week 8 | 0.58 (2.57)
  P-alb, Week 16: number analyzed (Participants) | 150
  P-alb, Week 16 | 1.18 (2.91)
  P-alb, Week 24: number analyzed (Participants) | 150
  P-alb, Week 24 | 1.4 (3.18)
  P-alb, Week 52: number analyzed (Participants) | 126
  P-alb, Week 52 | 1.83 (3.23)

48. Secondary Outcome: Change From Baseline in B-leuk, B-ly, B-neutr and B-Thromb Levels at Week 8, Week 16, Week 24 and Week 52
Description: Baseline was considered as date of initiation of tofacitinib.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
10^9 cells per liter
  B-leuk, Week 8: number analyzed (Participants) | 213
  B-leuk, Week 8 | -3.31 (33.44)
  B-leuk, Week 16: number analyzed (Participants) | 213
  B-leuk, Week 16 | -4.34 (36.02)
  B-leuk, Week 24: number analyzed (Participants) | 213
  B-leuk, Week 24 | -4.81 (38.2)
  B-leuk, Week 52: number analyzed (Participants) | 181
  B-leuk, Week 52 | -2.34 (3.12)
  B-ly, Week 8: number analyzed (Participants) | 149
  B-ly, Week 8 | 0.18 (0.86)
  B-ly, Week 16: number analyzed (Participants) | 149
  B-ly, Week 16 | 0.06 (0.81)
  B-ly, Week 24: number analyzed (Participants) | 149
  B-ly, Week 24 | -0.03 (0.85)
  B-ly, Week 52: number analyzed (Participants) | 124
  B-ly, Week 52 | -0.14 (0.73)
  B-neutr, Week 8: number analyzed (Participants) | 146
  B-neutr, Week 8 | -1.27 (3.48)
  B-neutr, Week 16: number analyzed (Participants) | 146
  B-neutr, Week 16 | -1.77 (4.37)
  B-neutr, Week 24: number analyzed (Participants) | 146
  B-neutr, Week 24 | -2.22 (4.38)
  B-neutr, Week 52: number analyzed (Participants) | 120
  B-neutr, Week 52 | -2.11 (3.43)
  B-Thromb, Week 8: number analyzed (Participants) | 210
  B-Thromb, Week 8 | -25.22 (77.73)
  B-Thromb, Week 16: number analyzed (Participants) | 210
  B-Thromb, Week 16 | -33.59 (93.49)
  B-Thromb, Week 24: number analyzed (Participants) | 210
  B-Thromb, Week 24 | -36.54 (99.47)
  B-Thromb, Week 52: number analyzed (Participants) | 178
  B-Thromb, Week 52 | -40.14 (68.13)

49. Secondary Outcome: Percentage of Participants With Extended Tofacitinib Induction Dose at Week 8, Week 16
Description: Percentage of participants with extended tofacitinib induction dose (additional 8 weeks with 10 mg) is presented in this outcome measure.
Time Frame: Week 8 and Week 16
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of participants
  Week 8: number analyzed (Participants) | 241
  Week 8 | 69.71
  Week 16: number analyzed (Participants) | 251
  Week 16 | 36.25

50. Secondary Outcome: Percentage of Participants With Higher Dose (10 mg) of Tofacitinib For All Participants at Week 8, Week 16, Week 24 and Week 52
Description: Percentage of participants with higher dose (10 mg) of tofacitinib (for all participants) is presented in this outcome measure.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Percentage of Participants
  Week 8: number analyzed (Participants) | 241
  Week 8 | 75.93
  Week 16: number analyzed (Participants) | 251
  Week 16 | 40.24
  Week 24: number analyzed (Participants) | 251
  Week 24 | 30.28
  Week 52: number analyzed (Participants) | 212
  Week 52 | 17.45

51. Secondary Outcome: Number of Participants With Higher Dose (10mg) of Tofacitinib of Those on Treatment at Week 8, Week 16, Week 24 and Week 52
Description: Percentage of participants with higher (10 mg) dose of tofacitinib in participants who received treatment at different timepoints is presented in this outcome measure.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  Week 8: number analyzed (Participants) | 241
  Week 8 | 183
  Week 16: number analyzed (Participants) | 251
  Week 16 | 101
  Week 24: number analyzed (Participants) | 251
  Week 24 | 76
  Week 52: number analyzed (Participants) | 212
  Week 52 | 37

52. Secondary Outcome: Time to Drug Discontinuation, Colectomy or UC-related Hospitalization
Description: Time to survival without drug discontinuation, colectomy or UC-related hospitalization was calculated using time to event analysis.
Time Frame: Up to Week 52
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Months | 14.3 [10 to 25]

53. Secondary Outcome: Number of Previous Treatments
Description: Number of previous treatments received by participants is presented in this outcome measure.
Time Frame: Up to Week 52
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Mean (Standard Deviation); unit: Treatments
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Treatments | 4.5 (1.3)

54. Secondary Outcome: Number of Participants According to Type of Previous Treatment
Description: Number of participants according to type of their previous treatment received is presented.
Time Frame: Up to Week 52
Population: All eligible participants for whom data was collected and analyzed were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  Corticosteroids | 229
  5-aminosalicylic acid | 237
  Tiopurines combined | 222
  Azathioprine | 182
  6-Mercaptopurine | 93
  Methotrexate | 23
  Ciclosporin | 21
  Ustekinumab | 19
  Vedolizumab | 85
  Adalimumab | 61
  Infliximab | 159
  Golimumab | 20
  Bio naïve | 48
  Bioexperienced | 204

55. Secondary Outcome: Number of Participants With Steroid-free Clinical Remission of Those Treated With Corticosteroids at Baseline Based on Full Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: Clinical remission in participants was defined as a full Mayo score of <=2 points, with no individual sub score exceeding 1 point with rectal bleeding sub-score of 0. Full Mayo score consisted of 4 sub scores: rectal bleeding, stool frequency, physician assessment of disease activity, and endoscopy findings, each graded from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). These sub scores were summed up to give a total score range of 0 to 12, where higher scores indicated higher disease severity. Steroid-free clinical remission was defined as participants who were treated with corticosteroids at baseline and did not require any corticosteroid treatment during the period >=4 weeks prior to the visit.
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  Week 8: number analyzed (Participants) | 173
  Week 8 | 0
  Week 16: number analyzed (Participants) | 177
  Week 16 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 24: number analyzed (Participants) | 186
  Week 24 | 6
  Week 52: number analyzed (Participants) | 174
  Week 52 | 11

56. Secondary Outcome: Number of Participants With Steroid-free Clinical Remission of Those Treated With Corticosteroids at Baseline Based on Partial Mayo Score at Week 8, Week 16, Week 24 and Week 52
Description: as for outcome 14
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Participants
  Week 8: number analyzed (Participants) | 240
  Week 8 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 16: number analyzed (Participants) | 241
  Week 16 | 36
  Week 24: number analyzed (Participants) | 241
  Week 24 | 32
  Week 52: number analyzed (Participants) | 207
  Week 52 | 32

57. Secondary Outcome: Percentage of Participants That Had f-Calprotectin Above 250 mg/kg at Baseline
Description: F-calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Percentage of Participants That had f-Calprotectin Above 250 mg/kg at Baseline is presented.
Time Frame: At index (date of initiation of tofacitinib treatment for ulcerative colitis)
Population: All eligible participants for whom data was collected and analyzed were included. 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 189
Percentage of Participants | 90.5

58. Secondary Outcome: Change From Baseline in F-calprotectin at Week 8, Week 16, Week 24 and Week 52
Description: as for outcome 20
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Milligrams per kilogram
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Milligrams per kilogram
  Week 8: number analyzed (Participants) | 189
  Week 8 | -511.55 (1281.31)
  Week 16: number analyzed (Participants) | 189
  Week 16 | -955.7 (1617.43)
  Week 24: number analyzed (Participants) | 189
  Week 24 | -1092.93 (1583.33)
  Week 52: number analyzed (Participants) | 158
  Week 52 | -1179.35 (1728.6)

59. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission for Those Treated With Corticosteroids at Baseline Based on Full Mayo Score From Week 16 to Week 24 and Week 52
Description: as for outcome 25
Time Frame: From Week 16 to Week 24 and Week 52
Population: as for outcome 32
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 4
Percentage of Participants
  Week 16 to Week 24 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.
  Week 16 to Week 52 | NA — Results having less than 5 participants with events could not be exported from the Finnish Health and Social Data Permit Authority (Findata) servers.

60. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission for Those Treated With Corticosteroids at Baseline Based on Partial Mayo Score From Week 16 to Week 24 and Week 52
Description: as for outcome 26
Time Frame: From Week 16 to Week 24 and Week 52
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 36
Percentage of Participants
  Week 16 to Week 24 | 63.89
  Week 16 to Week 52: number analyzed (Participants) | 29
  Week 16 to Week 52 | 44.83

61. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission for Those Treated With Corticosteroids at Baseline Based on Partial Mayo Score and Endoscopic Remission, Mucosal Healing or Endoscopic Response From Week 8 to Week 16, Week 24 and Week 52
Description: as for outcome 33
Time Frame: From Week 8 to Week 16, Week 24 and Week 52
Population: All eligible participants for whom data was collected and analyzed were included. Here, 'No participants fulfilled the criteria for the analysis'.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 0

62. Secondary Outcome: Percentage of Participants in Sustained Steroid Free Remission for Those Treated With Corticosteroids at Baseline Based on Full Mayo Score and Endoscopic Remission, Mucosal Healing or Endoscopic Response From Week 8 to Week 16, Week 24 and Week 52
Description: as for outcome 32
Time Frame: From Week 8 to Week 16, Week 24 and Week 52
Population: as for outcome 61
Arm/Group | Tofacitinib
Number analyzed (Participants) | 0

63. Secondary Outcome: Absolute Values of Blood Hemoglobin and Plasma Albumin at Baseline
Description: Absolute Values of Blood Hemoglobin and Plasma Albumin at Baseline are presented in this outcome measure.
Time Frame: At index (from data collected and analyzed retrospectively over 5 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 252
Grams per liter
  Blood hemoglobin (female): number analyzed (Participants) | 77
  Blood hemoglobin (female) | 126.73 (12.64)
  Blood hemoglobin (male): number analyzed (Participants) | 175
  Blood hemoglobin (male) | 139.22 (15.99)
  Plasma albumin: number analyzed (Participants) | 150
  Plasma albumin | 36.49 (4.28)

ADVERSE EVENTS:
Time Frame: Not applicable for this study as safety data was not planned to be collected during the study
Description: This study involved data that existed as structured data. In these data sources, individual participant data could not be retrieved/ validated, it was not possible to link (i.e., identify potential association between) particular product and medical event for any individual. Thus, minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) was not met. Hence safety data was not collected and reported.
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT05082428/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT05082428/SAP_001.pdf